CLINICAL TRIAL: NCT07303153
Title: Assessment of Quality of Life After Acute Mesenteric Ischemia
Acronym: EQVIMA-1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9481
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Mesenteric Ischemia
Keywords: Acute Mesenteric Ischemia; Quality of Life After Acute Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute mesenteric ischemia is a severe abdominal emergency associated with a poor prognosis. While numerous studies have been conducted on the incidence, outcomes, and risk factors of mesenteric ischemia, very few focus on the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years)
* Treated for mesenteric ischemia between 2010 and 2022 in the intensive care, cardiovascular, and digestive and vascular surgery departments of the Strasbourg University Hospitals

Exclusion Criteria:

* Chronic mesenteric ischemia or other non-ischemic intestinal vascular pathologies such as mechanical causes.
* Colonic ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years) treated for mesenteric ischemia in the Strasbourg University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Score of GIQLI (Gastrointestinal Quality of Life Index) | Up to 12 months
  The GIQLI quality of life score consists of 36 items:
  the higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - CHU de Strasbourg - France, Strasbourg, France